CLINICAL TRIAL: NCT06880614
Title: Effect of House Cricket Preload on Glycemic Response in Type 2 Diabetes Patients
Brief Title: Effect of Acute Protein Supplementation in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, JERRY VANLIN, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: LPK2203
Record Dates: First submitted 2025-03-14; First posted 2025-03-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test; Whey

STUDY DESIGN:
Intervention Model Description: Randomized, Cross over, Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): This arm will be given chicken-flavored soup without any supplements before conducting the oral glucose tolerance test
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour); Dietary Supplement: Placebo
- Whey (Active Comparator): This arm will be given chicken-flavored soup containing whey isolate powder before conducting the oral glucose tolerance test
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour); Dietary Supplement: Whey
- House Cricket (Experimental): This arm will be given chicken-flavored soup containing house cricket powder before conducting the oral glucose tolerance test
  Interventions: Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour); Dietary Supplement: House cricket

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance test (75g 2-hour) — The participants are required to drink a glucose solution containing 75 g of glucose dissolved in 250 mL of water
Dietary Supplement: Whey — Supplemented with whey protein isolate masked with a chicken-flavored soup
  Arms: Whey
Dietary Supplement: House cricket — Supplemented with house cricket powder masked with chicken-flavored soup
  Arms: House Cricket
Dietary Supplement: Placebo — Placebo consists of chicken-flavored soup without any supplement inside
  Arms: Placebo

SUMMARY:
The goal of this trial is to test the effect of house cricket (Acheta domesticus) preload on glycemic response in diabetic patients. The main question[s] it aims to answer are: whether house cricket powder could lower blood glucose spike and stimulate higher insulin response. Participants will consume either house cricket powder, whey protein isolate or placebo which will be mixed with a chicken-flavored soup. Participants fingers will be pricked for up to 2 hours.

Researcher will compare house cricket powder with placebo to see if the glycemic response is better in house cricket supplemented group.

Researcher will compare house cricket powder with whey protein isolate to see if both supplement induce comparable glycemic response.

DETAILED DESCRIPTION:
Participants blood will be collected at 8 time points:

Baseline 20 minutes after pre load 15 minutes after Oral Glucose Tolerance Test (OGTT) 30 minutes after OGTT 45 minutes after OGTT 60 minutes after OGTT 90 minutes after OGTT 120 minutes after OGTT

ELIGIBILITY:
Inclusion Criteria:

* Suffering from type 2 diabetes mellitus (HbA1c > 6.5%)
* Consume metformin for at least 6 months

Exclusion Criteria:

* Consume other type of anti-diabetic drugs
* Presenting any food allergy
* Recent surgery or infections that may affect oral glucose tolerance test
* Consume other drugs that may affect oral glucose tolerance test
* Not consuming any anti-diabetic drugs
* Pre-diabetes (HbA1c 5.7 - 6.4%)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 120 minutes
  Blood glucose concentration measured using glucometer. Participants fingers are pricked and using capillary tube, a drop of the blood is dripped in a test strip before inserted to a glucometer.

SECONDARY OUTCOMES:
Blood insulin | 120 minutes
  Blood sample is collected through a finger prick. The blood will be centrifuged to obtain the serum. Insulin serum concentration is then measured by using ELISA kits. The blood sample are treated following the kit guideline, and the insulin concentration are measured by comparing the light absorbance against a prepared standard.

CONTACTS AND LOCATIONS:
Overall Officials: Ashril Yusof, PhD, Principal Investigator — University of Malaya
Locations (1):
- Queen Elizabeth Hospital Kota Kinabalu, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clifton PM, Galbraith C, Coles L. Effect of a low dose whey/guar preload on glycemic control in people with type 2 diabetes--a randomised controlled trial. Nutr J. 2014 Oct 25;13:103. doi: 10.1186/1475-2891-13-103. PMID 25343850
- [Background] Oberoi A, Giezenaar C, Rigda RS, Horowitz M, Jones KL, Chapman I, Soenen S. Effects of co-ingesting glucose and whey protein on blood glucose, plasma insulin and glucagon concentrations, and gastric emptying, in older men with and without type 2 diabetes. Diabetes Obes Metab. 2023 May;25(5):1321-1330. doi: 10.1111/dom.14983. Epub 2023 Feb 22. PMID 36694303
- [Background] Jakubowicz D, Froy O, Ahren B, Boaz M, Landau Z, Bar-Dayan Y, Ganz T, Barnea M, Wainstein J. Incretin, insulinotropic and glucose-lowering effects of whey protein pre-load in type 2 diabetes: a randomised clinical trial. Diabetologia. 2014 Sep;57(9):1807-11. doi: 10.1007/s00125-014-3305-x. Epub 2014 Jul 10. PMID 25005331
- [Background] Dai J, Lov J, Martin-Arrowsmith PW, Gritsas A, Churchward-Venne TA. The acute effects of insect vs. beef-derived protein on postprandial plasma aminoacidemia, appetite hormones, appetite sensations, and energy intake in healthy young men. Eur J Clin Nutr. 2022 Nov;76(11):1548-1556. doi: 10.1038/s41430-022-01157-8. Epub 2022 May 10. PMID 35538144
- [Background] Kashima H, Uemoto S, Eguchi K, Endo MY, Miura A, Kobayashi T, Fukuba Y. Effect of soy protein isolate preload on postprandial glycemic control in healthy humans. Nutrition. 2016 Sep;32(9):965-9. doi: 10.1016/j.nut.2016.02.014. Epub 2016 Mar 8. PMID 27157469